CLINICAL TRIAL: NCT04489888
Title: A Phase 4, Single-arm, Open-label Clinical Study of Pembrolizumab (MK-3475) to Evaluate the Efficacy and Safety of MK-3475 Plus Carboplatin and Paclitaxel as First-line Treatment of Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma (KEYNOTE B10).
Brief Title: A Study of Pembrolizumab (MK-3475) Plus Carboplatin and Paclitaxel as First-line Treatment of Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma (MK-3475-B10/KEYNOTE B10)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-B10; MK-3475-B10 (Other: MSD)
Record Dates: First submitted 2020-07-27; First posted 2020-07-28 (Actual); Results first posted 2024-05-09 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Carboplatin + Paclitaxel (Experimental): Participants will receive pembrolizumab plus carboplatin plus paclitaxel. Pembrolizumab will be administered via intravenous (IV) infusion at a dose of 200 mg on Day 1 of each 21-day cycle for up to 35 cycles (up to ~2 years). Carboplatin will be administered via IV infusion at area under curve (AUC) 5 mg/mL/minute on Day 1 of each 21-day cycle for up to 6 cycles (up to ~4 months). At investigator's choice, paclitaxel will be administered via IV infusion at a dose of 100 mg/m^2 on Day 1 and Day 8 of each 21-day cycle for up to 6 cycles (up to ~4 months) or at a dose of 175 mg/m^2 on Day 1 of each 21-day cycle for up to 6 cycles (up to ~4 months).
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg IV infusion given on Day 1 of each 21-day cycle
  Other Names: MK-3475; KEYTRUDA®
Drug: Carboplatin — Carboplatin AUC 5 mg/mL/minute IV infusion given on Day 1 of each 21-day cycle
  Other Names: PARAPLATIN®
Drug: Paclitaxel — At investigator's choice, paclitaxel 100 mg/m^2 IV infusion given on Day 1 and Day 8 of each 21-day cycle or paclitaxel 175 mg/m^2 IV infusion given on Day 1 of each 21-day cycle
  Other Names: TAXOL®; ONXAL®

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of pembrolizumab combined with carboplatin and paclitaxel as first-line treatment in participants with recurrent/metastatic head and neck squamous cell carcinoma (R/M HNSCC). No statistical hypothesis will be tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically-confirmed diagnosis of R/M HNSCC that is considered incurable by local therapies
* Male participants refrain from donating sperm plus are abstinent from heterosexual intercourse or agree to use contraception during the intervention period and for at least 95 days after carboplatin/paclitaxel
* Female participants are not pregnant or breastfeeding and are either not a woman of child-bearing potential (WOCBP) or use a contraceptive method that is highly effective or are abstinent from heterosexual intercourse during the intervention period and for at least 120 days after pembrolizumab or 30 days after paclitaxel or 6 months after carboplatin whichever occurs last, and agree not to donate or freeze eggs during this period
* Has adequate organ function

Exclusion Criteria:

* Has disease that is suitable for local therapy administered with curative intent
* Has a life expectancy of less than 3 months and/or has rapidly progressive disease
* Has a diagnosed and/or treated additional malignancy within 5 years prior to allocation with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, curatively resected in situ cervical cancer and curatively resected in situ breast cancer
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a history of or current non-infectious pneumonitis/interstitial lung disease that requires steroids
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B or Hepatitis C virus infection
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (35):
- United States (14):
  - Yale-New Haven Hospital-Yale Cancer Center ( Site 0265), New Haven, Connecticut
  - Helen F. Graham Cancer Center & Research Institute ( Site 0214), Newark, Delaware
  - Baptist MD Anderson Cancer Center ( Site 0215), Jacksonville, Florida
  - Orlando Health, Inc. ( Site 0216), Orlando, Florida
  - Regions Hospital ( Site 0227), Saint Paul, Minnesota
  - Washington University School of Medicine ( Site 0240), St Louis, Missouri
  - Erie County Medical Center-Head & Neck Surgery and Plastic & Reconstructive Surgery ( Site 0268), Buffalo, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 0262), Mineola, New York
  - Novant Health Presbyterian ( Site 0261), Charlotte, North Carolina
  - Novant Health Forsyth Medical Center ( Site 0266), Winston-Salem, North Carolina
  - UPMC Hillman Cancer Center ( Site 0253), Pittsburgh, Pennsylvania
  - Abington Hospital - Asplundh Cancer Center ( Site 0229), Willow Grove, Pennsylvania
  - Charleston Oncology ( Site 0231), Charleston, South Carolina
  - Virginia Commonwealth University ( Site 0233), Richmond, Virginia
- Argentina (5):
  - Hospital Provincial del Centenario ( Site 0304), Rosario, Santa Fe Province
  - Centro Medico San Roque ( Site 0302), San Miguel de Tucumán, Tucumán Province
  - IDIM Instituto de Diagnostico e Investigaciones Metabolicas ( Site 0303), Buenos Aires
  - Fundación Respirar ( Site 0306), Buenos Aires
  - Instituto Medico Especializado Alexander Fleming ( Site 0301), Buenos Aires
- Australia (4):
  - Orange Health Services ( Site 0106), Orange, New South Wales
  - The Townsville Hospital ( Site 0105), Douglas, Queensland
  - Gold Coast University Hospital ( Site 0103), Southport, Queensland
  - St Vincents Hospital Melbourne ( Site 0101), Fitzroy, Victoria
- Brazil (7):
  - Centro Regional Integrado de Oncologia ( Site 0403), Fortaleza, Ceará
  - CETUS Hospital Dia Oncologia ( Site 0400), Belo Horizonte, Minas Gerais
  - Liga Norte Riograndense Contra o Cancer ( Site 0404), Natal, Rio Grande do Norte
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia ( Site 0406), Ijuí, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0402), São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia ( Site 0401), São Paulo
  - A.C. Camargo Cancer Center ( Site 0405), São Paulo
- Canada (5):
  - Tom Baker Cancer Center ( Site 0014), Calgary, Alberta
  - Dr. H. Bliss Murphy Cancer Centre ( Site 0001), St. John's, Newfoundland and Labrador
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital ( Site 0004), Kingston, Ontario
  - Princess Margaret Cancer Centre ( Site 0005), Toronto, Ontario
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 0003), Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Dzienis M, Cundom J, Fuentes CS, Spreafico A, Nordlinger M, Pastor AV, Alesi E, Neki A, Fung AS, Figueiredo Lima IP, Oppelt P, da Cunha Junior GF, Burtness B, Franke FA, Tseng JE, Joshi A, McCarthy J, Swaby R, Sidi Y, Gumuscu B, Naicker N, de Castro G Jr. Pembrolizumab Plus Carboplatin and Paclitaxel as First-Line Therapy for Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma (KEYNOTE-B10): A Single-Arm Phase IV Trial. J Clin Oncol. 2024 Sep 1;42(25):2989-2999. doi: 10.1200/JCO.23.02625. Epub 2024 Jul 22. PMID 39038265
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 101 participants were enrolled in the All Participants as Treated (APaT) population. The APaT population consisted of all allocated participants who received at least one dose of study intervention.
Groups:
- Pembrolizumab + Carboplatin + Paclitaxel: Participants received pembrolizumab plus carboplatin plus paclitaxel. Pembrolizumab was administered via intravenous (IV) infusion at a dose of 200 mg on Day 1 of each 21-day cycle for up to 35 cycles (up to ~2 years). Carboplatin was administered via IV infusion at area under curve (AUC) 5 mg/mL/minute on Day 1 of each 21-day cycle for up to 6 cycles (up to ~4 months). At investigator's choice, paclitaxel was administered via IV infusion at a dose of 100 mg/m^2 on Day 1 and Day 8 of each 21-day cycle for up to 6 cycles (up to ~4 months) or at a dose of 175 mg/m^2 on Day 1 of each 21-day cycle for up to 6 cycles (up to ~4 months).
Period: Overall Study
Arm/Group | Pembrolizumab + Carboplatin + Paclitaxel
Started | 101
Completed | 0
Not Completed | 101
Not completed — Death | 75
Not completed — Sponsor Decision | 26

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab + Carboplatin + Paclitaxel
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 88
  More than one race | 7
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters) per Response Evaluation Criteria in Solid Tumors Update and Clarification 1.1 (RECIST 1.1) which was adjusted for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The percentage of participants who experienced a CR or PR as assessed by blinded independent central review based on RECIST 1.1 was presented.
Time Frame: Up to ~25 months
Population: APaT population, which included all participants enrolled who received at least 1 dose of study intervention
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Carboplatin + Paclitaxel
Number analyzed (Participants) | 101
Percentage of Participants | 48.5 [38.4 to 58.7]

2. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrated a confirmed Complete Response (CR: Disappearance of all target lesions) or confirmed Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurred first. RECIST 1.1 was adjusted for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The DOR as assessed by blinded independent central review based on RECIST 1.1 was presented.
Time Frame: Up to ~25 months
Population: Participants in APaT population who had either a CR or PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Carboplatin + Paclitaxel
Number analyzed (Participants) | 49
Months | 5.5 [4.2 to 6.7]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from first dose of study treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. RECIST 1.1 was been adjusted for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ. PFS as assessed by blinded independent central review based on RECIST 1.1 was from product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to ~25 months
Population: APaT population, which included all participants enrolled who received at least 1 dose of study intervention
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Carboplatin + Paclitaxel
Number analyzed (Participants) | 101
Months | 5.6 [5.1 to 6.7]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of study treatment to death due to any cause. PFS as assessed by blinded independent central review based on RECIST 1.1 was from product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to ~25 months
Population: APaT population, which included all participants enrolled who received at least 1 dose of study intervention
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Carboplatin + Paclitaxel
Number analyzed (Participants) | 101
Months | 13.1 [9.6 to 15.2]

5. Secondary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced an AE was reported.
Time Frame: Up to ~39 months
Population: APaT population, which included all participants enrolled who received at least 1 dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Pembrolizumab + Carboplatin + Paclitaxel
Number analyzed (Participants) | 101
Percentage of participants | 100.0

6. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinued study treatment due to an AE was reported.
Time Frame: Up to ~25 months
Population: APaT population, which included all participants enrolled who received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pembrolizumab + Carboplatin + Paclitaxel
Number analyzed (Participants) | 101
Percentage of Participants | 36.6

ADVERSE EVENTS:
Time Frame: Up to approximately 39 months
Description: Serious and Other adverse events (AEs) include all participants who received ≥1 dose of study drug. All-Cause Mortality includes all allocated participants. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Data are reported by treatment received.
Arm/Group | Pembrolizumab + Carboplatin + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 75/101
Serious Adverse Events (participants affected / at risk) | 52/101
Other Adverse Events (participants affected / at risk) | 100/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Carboplatin + Paclitaxel (N=101)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6)
Atrial flutter (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Tongue necrosis (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Sudden death (General disorders) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 2 (2)
Endophthalmitis (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Infected fistula (Infections and infestations) | 1 (1)
Intestinal sepsis (Infections and infestations) | 1 (1)
Myelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 12 (13)
Pneumonia aspiration (Infections and infestations) | 6 (7)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (4)
Septic shock (Infections and infestations) | 2 (2)
Stoma site infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (5)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Vocal cord paralysis (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Carboplatin + Paclitaxel (N=101)
Anaemia (Blood and lymphatic system disorders) | 47 (64)
Ear pain (Ear and labyrinth disorders) | 6 (6)
Hypothyroidism (Endocrine disorders) | 19 (19)
Abdominal pain (Gastrointestinal disorders) | 11 (13)
Constipation (Gastrointestinal disorders) | 40 (57)
Diarrhoea (Gastrointestinal disorders) | 32 (64)
Dry mouth (Gastrointestinal disorders) | 13 (13)
Dyspepsia (Gastrointestinal disorders) | 9 (11)
Dysphagia (Gastrointestinal disorders) | 14 (14)
Nausea (Gastrointestinal disorders) | 36 (49)
Stomatitis (Gastrointestinal disorders) | 9 (11)
Vomiting (Gastrointestinal disorders) | 21 (31)
Asthenia (General disorders) | 13 (13)
Face oedema (General disorders) | 6 (6)
Fatigue (General disorders) | 47 (54)
Mucosal inflammation (General disorders) | 8 (9)
Oedema peripheral (General disorders) | 11 (11)
Pyrexia (General disorders) | 10 (11)
COVID-19 (Infections and infestations) | 7 (7)
Candida infection (Infections and infestations) | 6 (7)
Oral candidiasis (Infections and infestations) | 6 (7)
Pneumonia (Infections and infestations) | 15 (16)
Fall (Injury, poisoning and procedural complications) | 7 (8)
Alanine aminotransferase increased (Investigations) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 10 (10)
Blood alkaline phosphatase increased (Investigations) | 9 (13)
Blood creatinine increased (Investigations) | 11 (15)
Lymphocyte count decreased (Investigations) | 25 (44)
Neutrophil count decreased (Investigations) | 57 (140)
Platelet count decreased (Investigations) | 32 (63)
Weight decreased (Investigations) | 23 (25)
White blood cell count decreased (Investigations) | 34 (87)
Decreased appetite (Metabolism and nutrition disorders) | 25 (28)
Dehydration (Metabolism and nutrition disorders) | 12 (16)
Hypercalcaemia (Metabolism and nutrition disorders) | 8 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (16)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 (17)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (19)
Hypomagnesaemia (Metabolism and nutrition disorders) | 16 (20)
Hyponatraemia (Metabolism and nutrition disorders) | 15 (29)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (34)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (20)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (13)
Dizziness (Nervous system disorders) | 14 (16)
Dysgeusia (Nervous system disorders) | 11 (11)
Headache (Nervous system disorders) | 14 (21)
Neuropathy peripheral (Nervous system disorders) | 14 (14)
Paraesthesia (Nervous system disorders) | 11 (12)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (13)
Insomnia (Psychiatric disorders) | 15 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (18)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 35 (35)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (20)
Rash (Skin and subcutaneous tissue disorders) | 14 (20)
Hypertension (Vascular disorders) | 13 (29)
Hypotension (Vascular disorders) | 12 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity was not directed by the Sponsor, the investigator agreed to submit all manuscripts or abstracts to the Sponsor before submission. This allowed the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT04489888/Prot_SAP_002.pdf